CLINICAL TRIAL: NCT04439890
Title: A Randomized, Double-blind, Multicenter Phase III Study of Anlotinib Hydrochloride Capsule Combined With Chemotherapy Versus Placebo Combined With Chemotherapy as First-line Treatment in Subjects With Advanced Non-squamous Cell Non-small Cell Lung Cancer
Brief Title: A Efficacy and Safety Study of Anlotinib Hydrochloride Capsule Combined With Chemotherapy Versus Placebo Combined With Chemotherapy as First-line Treatment in Subjects With Advanced Non-squamous Cell Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-03-III-01
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Advanced Non-squamous Cell Non-small Cell Lung Cancer
MeSH Terms: interventions — Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib hydrochloride capsule + chemotherapy (Experimental): Anlotinib hydrochloride capsule 12mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) + Carboplatin injection (AUC 5mg/mL/min, intravenous drip, on Day 1) + Pemetrexed disodium f Injection (500mg / m2, intravenous drip, on Day 1).
  Interventions: Drug: Anlotinib hydrochloride capsule; Drug: Carboplatin injection; Drug: Pemetrexed disodium f Injection
- Placebo + chemotherapy (Placebo Comparator): Placebo given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) + Carboplatin injection (AUC 5mg/mL/min, intravenous drip, on Day 1) + Pemetrexed disodium f Injection (500mg / m2, intravenous drip, on Day 1).
  Interventions: Drug: Carboplatin injection; Drug: Pemetrexed disodium f Injection; Drug: Placebo

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsule — Anlotinib hydrochloride capsule 12mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Arms: Anlotinib hydrochloride capsule + chemotherapy
Drug: Carboplatin injection — Carboplatin injection AUC 5mg/mL/min, intravenous drip, on Day 1 in 21-day cycle.
Drug: Pemetrexed disodium f Injection — Pemetrexed disodium f Injection 500mg / m2, intravenous drip, on Day 1 in 21-day cycle.
Drug: Placebo — Placebo
  Arms: Placebo + chemotherapy

SUMMARY:
This is a randomized, double-blind, multicenter phase III clinical study to evaluate efficacy and safety of anlotinib hydrochloride capsule combined with chemotherapy versus placebo combined with chemotherapy as first-line treatment in subjects with advanced non-squamous cell non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Local advanced (stage IIIB / ⅢC), metastatic or recurrent (stage IV) non-squamous cell non-small cell lung cancer, has at least one measurable lesion.

  2. EGFR, ALK, and ROS1 test results are negative. 3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, life expectancy≥ 12 weeks.

  4. Has not received systemic anti-tumor treatment for advanced disease. 5.Adequate organ system function. 6. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ; No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

  7. Understood and signed an informed consent form.

Exclusion Criteria:

* 1.Other histopathological types of non-small cell lung cancer. 2.Has received VEGF pathway targeted therapy including anlotinib and bevacizumab.

  3. Has multiple factors affecting oral medication. 4. Has symptomatic brain metastases. 5. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.

  6. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1.

  7. Has any severe and / or uncontrolled diseases. 8. Has any bleeding symptoms or treated with anticoagulants or vitamin K antagonists.

  9.Has received surgery, or unhealed wounds within 4 weeks before the first administration.

  10. Has hemoptysis within 28 days before randomization. 11. Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear.

  12. Has arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident including transient ischemic attack, deep vein thrombosis and pulmonary embolism.

  13. Has psychotropic substances abuse or a mental disorder. 14. Have a history of immunodeficiency. 15. Has received allogeneic organ transplantation, hematopoietic stem cell transplantation or bone marrow transplantation.

  16. Has other malignancy. 17.Has participated in other anticancer drug clinical trials within 4 weeks. 18.According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to 48 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.

SECONDARY OUTCOMES:
Overall response rate (ORR) assessed by Independent Review Committee (IRC) | up to 48 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) based on IRC.
Overall survival (OS) | up to 48 weeks
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
Disease control rate（DCR） | up to 48 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Disease of Response (DOR) | up to 48 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (59):
- China (59):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Anhui Chest Hospital, Hefei, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Sixth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences, Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chinese PLA Army Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Wuwei Tumor Hospital, Wuwei, Gansu
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Huazhong University of Science Tongji Hospital, Tongji Medical College, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Changzhou Second People's Hospital, Changzhou, Jiangsu
  - Lianyungang First People's Hospital, Lianyungang, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Subei People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Neimenggu
  - Ningxia Medical University General Hospital, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Tengzhou Central People's Hospital, Tengzhou, Shandong
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tangdu Hospital, The Fourth Military Medical University of PLA, Xi’an, Shanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Dazhou Central Hospital, Dazhou, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ruian People's Hospital, Ruian, Zhejiang